CLINICAL TRIAL: NCT06005688
Title: An Interventional, Phase 1, Open-Label, Fixed Sequence, 2-Period Study to Estimate the Effect of Multiple Doses of Carbamazepine on the Pharmacokinetics of Single Dose Vepdegestrant (ARV-471, PF-07850327) 200 mg Under the Fed Condition in Healthy Adult Males and Females of Nonchildbearing Potential
Brief Title: A Study to Understand the Effects of Carbamazepine on How Vepdegestrant is Processed in Healthy Participants
Acronym: PK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Arvinas Estrogen Receptor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C4891011; 2023-505881-27 (EudraCT Number)
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Carbamazepine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vepdegestrant with and without Carbamazepine (Experimental): Vepdegestrant administered as a single dose in Period 1 and Period 2. Carbamazepine administered once a day for 19 days in Period 2.
  Interventions: Drug: Vepdegestrant; Drug: Carbamazepine

INTERVENTIONS:
Drug: Vepdegestrant — Participants will receive a single dose of Vepdegestrant by mouth in Period 1 and Period 2, with a washout period of at least 20 days between two doses of Vepdegestrant.
  Other Names: ARV-471, PF-07850327
Drug: Carbamazepine — Participants will receive Carbamazepine by mouth once a day for 19 days in Period 2.
  Other Names: Tegretol

SUMMARY:
The purpose of this study is to understand if carbamazepine reacts with vepdegestrant and affects how it is processed in the bodies of healthy participants.

This study is seeking participants who:

* are male, or female who cannot have children.
* are 18 years or older.
* are extremely healthy as decided by medical tests.
* have a body mass index (BMI) of 16 to 32 kilogram per meter squared.
* have a total body weight of more than 45 kilograms (99 pounds).
* can understand the study needs and provide a signed document to take part in the study.

All participants in this study will receive one dose of vepdegestrant alone by mouth in Period 1. In Period 2, all participants will receive carbamazepine by mouth once a day for 19 days. Participants will also receive one dose of vepdegestrant by mouth.

The levels of vepdegestrant in Period 1 will be compared to the levels of vepdegestrant in Period 2 to decide if carbamazepine affects how vepdegestrant is processed differently in healthy adults.

The study duration is 27 days and includes two periods. Participants will stay in the clinical research unit through the end of period 2. The participants may be allowed to leave on Day 4 or at the end of Period 1 but must return at the study doctor's call to complete the study. A follow-up visit for each participant takes place at 28 to 35 days after taking the study medicine for the last time.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants, and female participants of non-childbearing potential aged 18 years or older (or the minimum age of consent in accordance with local regulations) at screening who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
2. BMI of 16-32 kg/m2; and a total body weight >45 kg (99.2 lb).
3. Capable of giving signed informed consent, which includes compliance with requirements and restrictions listed in the ICD and in this protocol.
4. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

   * Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
   * History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, HBcAb, or HCVAb. Hepatitis B vaccination is allowed.
2. Participants shown to carry or be positive for HLA-B*1502 and/or HLA-A*3101 (genotyping alleles/markers related with carbamazepine-associated SJS or TEN).
3. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
4. Use of prescription or non-prescription medications, including vitamins, herbal and dietary supplements, grapefruit/grapefruit containing products, and Seville orange/Seville orange containing products within 7 days prior to the first dose of study intervention with the exception of:

   * Moderate/strong CYP3A4 inducers which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
   * Moderate/strong CYP3A4 inhibitors which are prohibited within 14 days plus 5 half-lives prior to the first dose of study intervention.
5. Previous administration with an investigational product (drug or vaccine) within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
6. A positive urine drug test. A single repeat for positive drug screen may be allowed.
7. Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic) for participants <60 years; and ≥150/90 mm Hg for participants ≥60 years old, following at least 5 minutes of supine rest. If systolic BP is ≥140 or 150 mm Hg (based on age) or diastolic ≥90 mm Hg, the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
8. Baseline standard 12-lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
9. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

   • AST, ALT, or Total Bilirubin Level >1.05× ULN;
10. Renal impairment as defined by an eGFR <60 mL/min/1.73m². Based upon participant age at screening, eGFR is calculated usding the recommended CKD-EPI equations to determine eligibility and to provide a baseline to quantify any subsequent kidney safety events.
11. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit, or 3 ounces (90 mL) of wine).
12. History of use of tobacco or nicotine-containing products in excess of the equivalent of 5 cigarettes/day or 2 chews of tobacco/day.
13. History of sensitivity to vepdegestrant and Tegretol or any of the formulation components of vepdegestrant and Tegretol.
14. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-08-18 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Vepdegestrant when administered alone | Period 1 - Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 144 hour post-dose
Cmax of Vepdegestrant when administered with carbamazepine | Period 2 - Day 14 pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 144 hour post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of Vepdegestrant when administered alone | Period 1 - Day 1 pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 144 hour post-dose
AUCinf of Vepdegestrant when administered with carbamazepine | Period 2 - Day 14 pre-dose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, and 144 hour post-dose

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Time the participant provides informed consent through and including follow-up contact occurring 28 to 35 calendar days after the last administration of the study intervention.
Number of Participants With Clinical Laboratory Abnormalities | Baseline up to Period 2 Day 20
Number of Participants With Electrocardiogram (ECG) Abnormalities | Baseline up to Period 2 Day 20
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to Period 2 Day 20
Number of Participants With Abnormalities in Physical Examinations | Baseline up to Period 2 Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4891011